CLINICAL TRIAL: NCT00730314
Title: Phase I/II Trial Of Hematopoietic Stem Cell Transplant (HSCT) For Children With A Genetic Disease Of Blood Cells Without An HLA-Matched Sibling Donor
Brief Title: Unrelated Hematopoietic Stem Cell Transplantation(HSCT) for Genetic Diseases of Blood Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Hisham Abdel-Azim, Principle Investigator, Children's Hospital Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCI #07-00119; CHLA-#07-00119
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Sickle Cell Disease; Thalassemia; Anemia; Granuloma; Wiskott-Aldrich Syndrome; Chediak Higashi Syndrome; Osteopetrosis; Neutropenia; Thrombocytopenia; Hurler Disease; Niemann-Pick Disease; Fucosidosis
Keywords: unrelated; BMT; HSCT; bone marrow transplantation; sickle cell disease; thalassemia; CGD; HLH; Blackfan-Diamond anemia; Hurler; leukodystrophy; LAD I; Genetic diseases; Red blood cell defects; Leukocyte defects and immune deficiencies; Hereditary Lymphohistiocytosis; chronic granulomatous disease; Wiskott-Aldrich syndrome; Chediak Higashi syndrome; CD40 ligand deficiency; Hyper IgM syndrome; leucocytes adhesion defect type 1; Osteopetrosis; congenital neutropenia; X-linked lymphoproliferative disease; Platelets defects; Congenital amegakaryocytic thrombocytopenia; Metabolic and storage disorders; Hurler disease; leukodystrophies; Niemann-Pick disease; Fucosidosis; Stem cell defects; reticular agenesis
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Anemia; Granuloma; Wiskott-Aldrich Syndrome; Chediak-Higashi Syndrome; Osteopetrosis; Neutropenia; Thrombocytopenia; Mucopolysaccharidosis I; Niemann-Pick Diseases; Fucosidosis; Anemia, Dyserythropoietic, Congenital; Genetic Diseases, Inborn; Granulomatous Disease, Chronic; Hyper-IgM Immunodeficiency Syndrome; Neutropenia, Severe Congenital, Autosomal Recessive 3; Lymphoproliferative Disorders; Congenital amegakaryocytic thrombocytopenia | interventions — Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Unrelated donor
  Interventions: Procedure: Hematopoietic stem cell transplantation
- 2 (Experimental): Cord Blood
  Interventions: Procedure: Hematopoietic stem cell transplantation

INTERVENTIONS:
Procedure: Hematopoietic stem cell transplantation — hematopoietic stem cell transplantation conditioning regimen depending on graft source

SUMMARY:
This is a clinical trial of bone marrow transplantation for patients with the diagnosis of a genetic disease of blood cells that do not have an HLA-matched sibling donor. Genetic diseases of blood cell include: Red blood cell defects e.g. hemoglobinopathies (sickle cell disease and thalassemia), Blackfan-Diamond anemia and congenital or chronic hemolytic anemias; White blood cells defects/immune deficiencies e.g. chronic granulomatous disease, Wiskott-Aldrich syndrome,Osteopetrosis, Kostmann's syndrome (congenital neutropenia), Hereditary Lymphohistiocytosis (HLH); Platelets defects e.g.Congenital amegakaryocytic thrombocytopenia; Metabolic/storage disorders e.g. leukodystrophies,mucopolysaccharidoses as Hurler disease;Stem cell defects e.g.reticular agenesis, among many other rare similar conditions.

The study treatment plan uses a new transplant treatment regimen that aims to try to decrease the acute toxicities and complications associated with the standard treatment plans and to improve outcome

The blood stem cells will be derived from either unrelated donor or unrelated umbilical cord blood.

DETAILED DESCRIPTION:
This is a pilot clinical trial of hematopoietic stem cell transplantation for patients with the diagnosis of a genetic disease of blood cells that do not have an HLA-matched sibling donor. The stem cells will be derived from a 1) matched unrelated donor (MUD) or 2) unrelated umbilical cord blood (UCB). Patients will receive a novel conditioning regimen with Busulfan, Cytoxan and Fludarabine (Bu/Cy/Flu) and either Alemtuzumab (Campath 1H) for recipients of a MUD or rabbit Antithymocyte Globulin (rATG) for recipients of unrelated UCB prior to hematopoietic stem cell transplant (HSCT).

It is hypothesized that reduced dosages of Cytoxan will decrease the acute toxicities associated with the standard chemotherapies of Busulfan and Cytoxan (i.e. sinusoidal obstructive syndrome (SOS), hemorrhagic cystitis and mucositis). And the addition of fludarabine to a conditioning regimen with myeloablative doses of Busulfan and reduced dosages of Cytoxan prior to HSCT will overcome the engraftment barrier posed by an intact immune system, which is seen in patients with a genetic disease.

ELIGIBILITY:
Inclusion Criteria:

* Lethal or sublethal genetic disease of blood cells, who lack a fully histocompatible sibling or other family donor
* Genetic diseases that would be candidates for this protocol includes those that have been shown to benefit from allogeneic HSCT: Red blood cell defects, Leukocyte defects/ Primary immune deficiencies, Platelets defects, Metabolic/storage disorders and Stem cell defects.
* Renal: creatinine clearance or glomerular filtration rate (GFR) ≥50 ml/min/1.73m2 and not requiring dialysis.
* Pulmonary: FEV1, FVC and DLCO (corrected for hemoglobin) ≥ 50% predicted. if unable to perform pulmonary function tests, then O2 saturation ≥ 92% in room air.
* Cardiac: Left ventricular ejection fraction at rest must be ≥ 40%, or shortening fraction ≥ 26%
* Hepatic: Bilirubin ≤3x upper limit of normal (ULN) and ALT and AST ≤ 5x for age (with the exception of isolated hyperbilirubinemia due to Gilbert's syndrome).
* Patients will be 0-21 years of age.
* Disease specific inclusion criteria (as applicable per protocol).

Exclusion Criteria:

* Recipients should not have any of the general exclusion criteria, and disease specific exclusion criteria when applicable.
* Patient with histocompatible sibling
* End-organ failure that precludes the ability to tolerate the transplant procedure, including the conditioning regimen.
* Creatinine clearance or GFR < 50 ml/min/1.73m2 or renal failure requiring dialysis.
* Congenital heart disease resulting in congestive heart failure.
* Severe residual CNS disease/impairment [(other than hemiplegia alone) e.g. coma or intractable seizures]
* Ventilatory failure
* Major congenital anomalies that adversely affect survival, e.g. CNS malformations
* Lansky score < 40% or Karnofsky score < 60%
* HIV seropositivity
* Diagnosis of Fanconi's anemia, Severe Combined Immunodeficiency (SCID)
* Positive pregnancy test (For female patients in child bearing period)
* Uncontrolled bacterial, viral, or fungal infections (currently taking medication yet clinical symptoms progress)
* Disease specific exclusion criteria (as applicable per protocol).

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2008-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
toxicities | 3 years
adverse events | 3 years
engraftment | 1 year
immune reconstitution | 3 years
overall and event free survival survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Abdel-Azim, MD, Principal Investigator — Childrens Hospital Los Angeles, University of Southern California
Locations (1):
- Children Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No